CLINICAL TRIAL: NCT03916796
Title: Rehabilitation and Quality of Life Assessment for Soft Tissue Sarcoma Treated With Radiotherapy and Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too many barriers to enrolling well going forward
Sponsor: Washington University School of Medicine (Other)
Collaborators: ReVital Cancer Rehabilitation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201904042
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Exercise; Enhanced Recovery After Surgery; Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Operative Radiotherapy: Dietary Counseling/Exercise/Psychological Counsel (Experimental): * Patients must be treated using daily image-guided radiotherapy
  * Dietary counseling at baseline
  * Exercise intervention throughout cancer rehabilitation protocol
  * Psychological screening with counselling services as needed - nurse will administer the NCCN distress thermometer and refer the patient to applicable psychological counselling
  Interventions: Other: Exercise; Other: Enhanced Recovery after surgery; Other: Psychological screening with counselling services as needed; Other: Dietary Counseling Services
- Post-Operative Radiotherapy: Dietary Counseling/Exercise/Psychological Counsel (Experimental): * Patients must be treated using daily image-guided radiotherapy
  * Dietary counseling at baseline
  * Exercise intervention throughout cancer rehabilitation protocol
  * Psychological screening with counselling services as needed - nurse will administer the NCCN distress thermometer and refer the patient to applicable psychological counselling
  Interventions: Other: Exercise; Other: Enhanced Recovery after surgery; Other: Psychological screening with counselling services as needed; Other: Dietary Counseling Services

INTERVENTIONS:
Other: Exercise — -The exercise part will consist of an evaluation and treatment as prescribed by a physical therapist including aerobic & dynamic stretching warm-up, strength training, balance training, and flexibility training. Will also include a home exercise program (HEP). Physical therapists will have specialized training in cancer rehabilitation obtained through the ReVital certification process.
Other: Enhanced Recovery after surgery — -The protocols include instructions for patient care from the time of pre-surgical admission to discharge, including directives regarding diet, labs, IV fluids, pain management, prophylactic medications, management of indwelling catheters and drains, and activity.
  Other Names: ERAS
Other: Psychological screening with counselling services as needed — -The psychological screening will be completed by the Radiation Oncology nurse at the consult visit
Other: Dietary Counseling Services — -Patients will have a baseline nutrition counseling visit with a Registered Dietician. This may include a nutrition assessment and nutrition counseling to set priorities, establish goals, and create an individualized plan

SUMMARY:
This is a pilot study with a feasibility lead-in evaluating the use of multimodal cancer rehabilitation in patients planning to undergo radiotherapy and surgical resection for extremity or superficial trunk soft tissue sarcoma (STS). At enrollment, patients will be assigned to either a pre-operative radiation or post-operative radiation cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft tissue sarcoma of the extremity, or superficial trunk (abdomen or chest)
* Planning to receive radiotherapy and surgical resection
* At least 16 years of age.
* ECOG performance status ≤ 3
* Able to complete the cancer rehabilitation protocol safely, as determined by a treating physician.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Patients deemed ineligible for curative therapy by the treating medical oncologist, radiation oncologist, or surgeon.
* Patients with deep retroperitoneal or abdominal STS
* Patients who have received prior radiotherapy and, based on the treating radiation oncologist's opinion, may not safely be treated with protocol neoadjuvant radiotherapy.
* Currently receiving any investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test prior to starting radiotherapy.
* HIV-positive patients whose CD4+ T-cell count is < 350 cells/mcL.
* Receiving concurrent chemoradiation therapy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Percentage of prescribed dietary and physical therapy visits completed during the cancer rehabilitation protocol | Through 3 month follow-up
  * This will be quantified as the proportion of prescribed visits within the prehabilitation protocol that are attended by the patient. If a patient participates in any portion of a prescribed visit, it will be counted as attended.
  * Physical therapy visits are optional from 6 months-24 months

SECONDARY OUTCOMES:
Rate of acute treatment-related grade 2 or higher toxicity attributed to the therapy | From baseline through 24 month follow-up
Quality of life as measured by the PROMIS Global total score | Change from baseline through 24 month follow-up
  -PROMIS scales to be used: Physical Function-10, Ability to Participate in Social Roles, Pain Interference, Anxiety and Depression, and Activities-4 and Global Health assessments. These are validated instruments with items ranked on a 5-point Likert scale. PROMIS is scored using T scores, which are standardized to the U.S. general population and have a mean of 50 and a standard deviation of 10. Scores above or below 50 are above or below the population average in the U.S. general population, respectively. The total T score will be calculated for this outcome measure
Quality of life as measured by the TESS | Change from baseline through 24 month follow-up
  -The Toronto Extremity Salvage Score was developed as a measure of patient reported physical functioning for patients undergoing limb salvage surgery for bone and STS
Patient cardiovascular capacity as measured by the 6-minute walk test | Change from baseline through 3 month follow-up
  -This test measures number of meters participants are able to walk in a level setting.
Patient general physical health status as measured by 30-second sit to stand test | Change from baseline through 3 month follow-up
  -The 30 second chair stand test is used to measure functional lower extremity strength and overall endurance. Participants are asked to go from a sitting position to standing from a chair as many times as they can within 30 seconds. Higher numbers of sit to stand correlate with increased physical function and lower body strength
Patient fall risk as measured by Timed Up and Go test | Change from baseline through 3 month follow-up
  -The Timed Up and Go is a performance test of physical mobility and fall risk. The TUG measures how long it takes the patient, in seconds, to stand up from a standard arm chair, walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down again. Scores of 11 or below are predictive of fall risk
Patient general physical health status as measured hand grip strength | Change from baseline through 3 month follow-up
  -Hand grip strength is measured with the Jamar hydraulic handgrip dynamometer. Measurement is completed with participant in seated position, holding arm at side, elbow at 90 degrees, and with dynamometer at either second or third position (based on size of hands, smaller hands position 2, larger hands position 3) and participants are encouraged to squeeze as much as possible, 3 times with a minute in between each trial. Number of pounds strength is recorded along with hand dominance. This measure is used to record upper body strength
Quality of life as measured by the Work Ability Index | Change from baseline through 24 month follow-up
  -This patient-reported outcome measure asks ability to work on a scale of 0-10 with 0 being unable, and 10 fully able. It follows with two items asking about reduction in physical and mental work ability due to cancer and its treatment. Lastly, it asks how many days the participant has been off work. For this assessment higher scores indicate better levels of work ability
Quality of life as measured by the history of previous falls | Change from baseline through 24 month follow-up
  -Asking patients to report the number of times they've fallen. Patients who respond they have fallen in the past is correlated to risk of treatment toxicity and risk of future falls
Acute wound complication rate | Within first 90 days following surgery
  -Wound complications include secondary procedures, deep wound packing, readmission to the hospital, wet dressings >4 weeks, or extended dressings >6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Spraker, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu